CLINICAL TRIAL: NCT00122109
Title: Telemedicine and Anger Management Groups for PTSD Veterans in the Hawaiian Islands
Brief Title: Telemedicine and Anger Management Groups With PTSD Veterans in the Hawaiian Islands
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TEL 03-080
Record Dates: First submitted 2005-07-18; First posted 2005-07-21 (Estimated); Results first posted 2014-10-16 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2014-08

CONDITIONS: Posttraumatic Stress Disorder
Keywords: Posttraumatic Stress Disorder; Anger Management; Telemedicine modality
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Videoteleconferencing AMT (Experimental): The experimental arm is the group condition that received the AMT treatment intervention via a videoteleconferencing modality as compared to the control condition which is the traditional face-to-face modality.
  Behavioral: 12 sessions Anger Management Therapy. Anger Management Treatment (AMT), a 12-session manual-driven cognitive-behavioral intervention developed and found efficacious for anger management treatment with substance abuse veterans and has been applied to the PTSD population. AMT is highly structured with both psychoeducational and psychotherapy components. AMT is aimed at reducing anger affect and aggression through increasing anger management skills.
  Interventions: Behavioral: 12 sessions Anger Management Therapy.
- Face to Face AMT (Active Comparator): The control arm is the group condition that received the AMT treatment intervention via a traditional face-to-face modality as compared to the experimental condition which is the videoteleconferencing modality.
  Behavioral: 12 sessions Anger Management Therapy. Anger Management Treatment (AMT), a 12-session manual-driven cognitive-behavioral intervention developed and found efficacious for anger management treatment with substance abuse veterans and has been applied to the PTSD population. AMT is highly structured with both psychoeducational and psychotherapy components. AMT is aimed at reducing anger affect and aggression through increasing anger management skills.
  Interventions: Behavioral: 12 sessions Anger Management Therapy.

INTERVENTIONS:
Behavioral: 12 sessions Anger Management Therapy. — Anger Management Treatment (AMT), a 12-session manual-driven cognitive-behavioral intervention developed and found efficacious for anger management treatment with substance abuse veterans and has been applied to the PTSD population. AMT is highly structured with both psychoeducational and psychotherapy components. AMT is aimed at reducing anger affect and aggression through increasing anger management skills.
  Other Names: AMT

SUMMARY:
Telemedicine has the potential to profoundly influence the delivery of specialized care to the remote veteran population suffering with PTSD. Preliminary research supports telemedicine technology as a possible solution to improve access to mental health services for veterans with PTSD. The proposed research is a treatment-outcome study that will assess the clinical efficacy of conducting an Anger Management Therapy (AMT) group treatment intervention using a videoteleconferencing (VTC) modality as compared to the traditional in-person modality with veterans who have PTSD and reside in remote locations on the Hawaiian Islands. AMT is a manual-guided cognitive-behavioral, skill based group intervention that has been used nationwide in VA substance abuse programs and most recently has been adopted by many VA PTSD Clinical Teams to treat anger-related to the sequelae of PTSD.

DETAILED DESCRIPTION:
Background: Posttraumatic stress disorder (PTSD) is a prevalent problem among military troops. Recovery from combat-related PTSD is often complicated by problems with anger. Veterans with difficulties managing PTSD-related anger may be particularly likely to live in remote geographical regions where access to specialized mental health care is often limited. Telemental health (TMH) has been touted as a potential means of increasing access to care in rural or remote areas. Objectives: This study compared the effectiveness of group Anger Management Therapy (AMT) delivered via videoteleconferencing (VTC) and in-person delivery in a sample of rural combat veterans with PTSD. The long-range objective of this project was to develop an empirically sound TMH protocol that will facilitate the extension of manual guided clinical services to remote sites via VTC. We hypothesized that providing a manualized group therapy intervention via VTC would result in similar reductions in anger symptoms as obtained from traditional in-person care. Further, we hypothesized that key process indicators (i.e., attrition, adherence, satisfaction, and therapeutic alliance) would not be significantly different between the VTC and in-person conditions. The specific objectives of this project were to: a) determine if group AMT delivered via VTC is as effective as the same intervention delivered in-person on clinical outcomes measuring reductions in anger symptoms and b) determine if group AMT delivered via VTC is as effective as the same intervention delivered in-person on group process outcomes. Methods: A randomized controlled non-inferiority trial of 125 male veterans with PTSD and anger difficulties was conducted at three Department of Veterans Affairs' outpatient clinics. Participants were randomly assigned to receive AMT delivered in a group setting with the therapist either in-person (N= 64) or via VTC (N= 61). Participants were assessed at baseline, mid-treatment, post-treatment, and 3 and 6-months post-treatment. The primary clinical outcome was reduction of anger difficulties, as measured by the Anger Expression and Trait Anger subscales of the State-Trait Anger Expression Inventory (STAXI-2) and the Novaco Anger Total Scale (NAS). Process variables were measured to assess the feasibility of AMT delivered via VTC. SAS MEANS procedure was used to calculate means and standard deviations for change from baseline at subsequent assessment points for both intent-to-treat and per-protocol analysis.

ELIGIBILITY:
Inclusion Criteria:

* male
* PTSD diagnosis
* anger level at Staxi Trait Score=22 or higher
* stable medication regime

Exclusion Criteria:

* current substance dependence
* current psychosis
* suicidal
* homicidal
* cognitive impairment

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2005-08; Primary Completion 2008-10 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leslie A Morland, PsyD, Principal Investigator — VA Pacific Islands Health Care System, Honolulu, HI
Locations (1):
- VA Pacific Islands Health Care System, Honolulu, HI, Honolulu, Hawaii, United States

REFERENCES:
- [Result] Greene CJ, Morland LA, Durkalski VL, Frueh BC. Noninferiority and equivalence designs: issues and implications for mental health research. J Trauma Stress. 2008 Oct;21(5):433-9. doi: 10.1002/jts.20367. PMID 18956449
- [Result] Greene CJ, Morland LA, Macdonald A, Frueh BC, Grubbs KM, Rosen CS. How does tele-mental health affect group therapy process? Secondary analysis of a noninferiority trial. J Consult Clin Psychol. 2010 Oct;78(5):746-50. doi: 10.1037/a0020158. PMID 20873910
- [Result] Morland LA, Greene CJ, Rosen CS, Foy D, Reilly P, Shore J, He Q, Frueh BC. Telemedicine for anger management therapy in a rural population of combat veterans with posttraumatic stress disorder: a randomized noninferiority trial. J Clin Psychiatry. 2010 Jul;71(7):855-63. doi: 10.4088/JCP.09m05604blu. Epub 2010 Jan 26. PMID 20122374
- [Result] Gros DF, Gros K, Acierno R, Frueh BC, Moreland L. Relation between treatment satisfaction and treatment outcome in veterans with posttraumatic stress disorder. Journal of psychopathology and behavioral assessment. 2013 Jun 28; 35(4):522-30.
- [Result] Macdonald A, Greene CJ, Torres JG, Frueh BC, Morland LA. Concordance between clinician-assessed and self-report ratings of posttraumatic stress disorder across three ethnoracial groups. Psychological trauma : theory, research, practice and policy. 2012 Jan 1; 24:doi: 10.1037/a0027313.
- [Result] Morland LA, Greene CJ, Grubbs K, Kloezeman K, Mackintosh MA, Rosen C, Frueh BC. Therapist adherence to manualized cognitive-behavioral therapy for anger management delivered to veterans with PTSD via videoconferencing. J Clin Psychol. 2011 Jun;67(6):629-38. doi: 10.1002/jclp.20779. Epub 2011 Feb 25. PMID 21360528
- [Result] Mackintosh MA, Morland LA, Kloezeman K, Greene CJ, Rosen CS, Elhai JD, Frueh BC. Predictors of anger treatment outcomes. J Clin Psychol. 2014 Oct;70(10):905-13. doi: 10.1002/jclp.22095. Epub 2014 Apr 17. PMID 24752837
- [Result] Morland LA, Raab M, Mackintosh MA, Rosen CS, Dismuke CE, Greene CJ, Frueh BC. Telemedicine: a cost-reducing means of delivering psychotherapy to rural combat veterans with PTSD. Telemed J E Health. 2013 Oct;19(10):754-9. doi: 10.1089/tmj.2012.0298. Epub 2013 Aug 9. PMID 23931729
- See also: National Center for PTSD provides and comprehensive information on the assessment, treatment, and epidemiology of Posttraumatic stress disorder — http://www.ptsd.va.gov/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment took place between 2005-2008. Participants were recruited across three VA Pacific Island Healthcare System clinical sites and Vet Centers across the Hawaiian Islands, Maui, and Oahu. Attempts were made to recruit 16 participants for each of 9 cohorts with 10 participants randomized into each conditon (VTC vs NP) within a cohort.
Pre-assignment Details: Of the 125 veterans who entered treatment, 112 attended at least 9 of 12 treatment sessions and were included in our completer sample (NP = 57 and VTC = 55).
Groups:
- Videoteleconferencing AMT: The experimental arm is the group condition that received the CPT treatment intervention via a videoteleconferencing modality as compared to the control condition which is the traditional face-to-face modality.
  Anger Management Therapy (AMT) group treatment intervention: 12-session CBT Anger Management Treatment conducted over a videoteleconferencing modality.
- Face to Face AMT: The control arm is the group condition that received the CPT treatment intervention face-to-face traditional modality as compared to the experimental condition which is the via a videoteleconferencing modality .
  Anger Management Therapy (AMT) group treatment intervention: 12-session CBT Anger Management Treatment conducted over a videoteleconferencing modality.
Period: Overall Study
Arm/Group | Videoteleconferencing AMT | Face to Face AMT
Started | 61 (ITT) | 64 (ITT)
Completed | 55 | 57
Not Completed | 6 | 7
Not completed — Did not meet criteria | 6 | 7

BASELINE CHARACTERISTICS:
Groups:
- Face to Face AMT: The control arm is the group condition that received the CPT treatment intervention via a traditional face to face modality as compared to the experimental condition which is the videoteleconferncing modality.
  Anger Management Therapy (AMT) group treatment intervention: 12-session CBT Anger Management Treatment conducted over a face to face modality.
- Total: Total of all reporting groups
Arm/Group | Videoteleconferencing AMT | Face to Face AMT | Total
Number analyzed (Participants) | 61 | 64 | 125
Age, Continuous [Mean (Full Range); unit: years] | 54.8 [24 to 80] | 54.6 [22 to 75] | 54.7 [22 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 61 | 64 | 125
Region of Enrollment [Number; unit: participants]
  United States | 61 | 64 | 125

OUTCOME MEASURES:

1. Primary Outcome: State-Trait Anger Inventory (STAXI-2) Anger Expression Index
Description: Anger expression was measured using the STAXI-2's 32-item Anger Expression Index (range 0 - 96). The STAXI-2 subscale have robust psychometric properties including high internal consistency, external validity, and construct validity. The Anger Expression Index provides a general measure of anger expression; assessing one's experience, expression and efforts to control anger. Higher scores indicate more problematic levels of anger and its expression.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Videoteleconferencing AMT: The experimental arm is the group condition that received the AMT treatment intervention via a videoteleconferencing modality as compared to the control condition which is the traditional face-to-face modality.
- Face to Face AMT: The control arm is the group condition that received the AMT treatment intervention via a traditional face-to-face modality as compared to the experimental condition which is the videoteleconferencing modality.
Arm/Group | Videoteleconferencing AMT | Face to Face AMT
Number analyzed (Participants) | 61 | 64
units on a scale | 56.7 (12.0) | 55.0 (10.3)

2. Primary Outcome: State-Trait Anger Inventory (STAXI-2) Anger Expression Subscale
Description: as for outcome 1
Time Frame: Post-treatment (2 weeks following last treatment session)
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Face to Face AMT: The control arm is the group condition that received the CPT treatment intervention via the traditional face to face modality as compared to the control condition which is the experimental videoteleconferencing modality.
  Anger Management Therapy (AMT) group treatment intervention: 12-session CBT Anger Management Treatment conducted over a videoteleconferencing modality.
Arm/Group | Videoteleconferencing AMT | Face to Face AMT
Number analyzed (Participants) | 61 | 64
units on a scale | 42.4 (16.2) | 46.6 (12.2)

3. Secondary Outcome: PTSD Checklist-military Version (PCL-M)
Description: Self report that measures severity of PTSD symptoms. The PCL-M measures the 17 cardinal symptoms of PTSD as described in the DSM-IV-TR. The scale ranges from 0 - 85 with higher scores indicating worse PTSD symptoms. PTSD symptoms were measured at baseline and post-treatment only.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Videoteleconferencing AMT | Face to Face AMT
Number analyzed (Participants) | 61 | 64
units on a scale | 64.5 (11.6) | 65.8 (10.8)

4. Primary Outcome: State-Trait Anger Inventory (STAXI-2) Anger Expression Subscale
Description: as for outcome 1
Time Frame: 3-month Follow Up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Videoteleconferencing AMT | Face to Face AMT
Number analyzed (Participants) | 61 | 64
units on a scale | 41.8 (15.3) | 47.0 (13.4)

5. Primary Outcome: State-Trait Anger Inventory (STAXI-2) Anger Expression Subscale
Description: as for outcome 1
Time Frame: 6-month Follow Up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Videoteleconferencing AMT | Face to Face AMT
Number analyzed (Participants) | 61 | 64
units on a scale | 42.0 (15.6) | 46.6 (15.3)

6. Primary Outcome: Novaco Anger Scale (NAS)
Description: Anger disposition was assessed using the total scale score from the Novaco Anger Scale. This 60-item measure (range = 60 - 180) is a well validated self-report instrument designed to measure cognitive, arousal, and behavioral aspects of anger in both clinical and non-patient populations. Higher scores indicate more anger-related symptoms.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Videoteleconferencing AMT | Face to Face AMT
Number analyzed (Participants) | 61 | 64
units on a scale | 109.3 (16.1) | 109.8 (14.0)

7. Primary Outcome: Novaco Anger Scale (NAS)
Description: as for outcome 6
Time Frame: Post-treatment (2 weeks following last treatment session)
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Face to Face AMT: The control arm is the group condition that received the CPT treatment intervention via a traditional face to face modality as compared to the experimental condition which is the videoteleconferencing modality.
  Anger Management Therapy (AMT) group treatment intervention: 12-session CBT Anger Management Treatment conducted over a face to face modality.
Arm/Group | Videoteleconferencing AMT | Face to Face AMT
Number analyzed (Participants) | 61 | 64
units on a scale | 94.2 (19.1) | 99.2 (17.1)

8. Primary Outcome: Novaco Anger Scale (NAS)
Description: as for outcome 6
Time Frame: 3-Month Follow Up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Videoteleconferencing AMT | Face to Face AMT
Number analyzed (Participants) | 61 | 64
units on a scale | 96.4 (18.4) | 105.2 (19.2)

9. Primary Outcome: Novaco Anger Scale (NAS)
Description: as for outcome 6
Time Frame: 6-Month Follow Up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Videoteleconferencing AMT | Face to Face AMT
Number analyzed (Participants) | 61 | 64
units on a scale | 97.7 (20.2) | 101.0 (22.5)

10. Secondary Outcome: PTSD Checklist-military Version (PCL-M)
Description: as for outcome 3
Time Frame: Post-treatment (2 weeks following last treatment session)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Videoteleconferencing AMT | Face to Face AMT
Number analyzed (Participants) | 61 | 64
units on a scale | 59.2 (15.0) | 57.4 (16.0)

ADVERSE EVENTS:
Time Frame: Throughout the duration of the assessment and intervention, up to 9 months
Groups:
- Videoteleconferencing AMT: The experimental arm is the group condition that received the AMT treatment intervention via a videoteleconferencing modality as compared to the control condition which is the traditional face-to-face modality.
  Anger Management Therapy (AMT) group treatment intervention: 12-session CBT Anger Management Treatment conducted over a videoteleconferencing modality.
- Face to Face AMT: The control arm is the group condition that received the AMT treatment intervention via a traditional face-to-face modality as compared to the experimental condition which is the videoteleconferencing modality.
  Anger Management Therapy (AMT) group treatment intervention: 12-session CBT Anger Management Treatment conducted over a videoteleconferencing modality.
Arm/Group | Videoteleconferencing AMT | Face to Face AMT
Serious Adverse Events (participants affected / at risk) | 0/61 | 0/64
Other Adverse Events (participants affected / at risk) | 0/61 | 0/64

LIMITATIONS AND CAVEATS:
We conservatively excluced participants with acute safety concerns (homicidal or suicidal) and current substance dependence. However other literature suugests that both issues can be safely addressed via telemedicine.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes